CLINICAL TRIAL: NCT06762977
Title: A Composite Assay for HER2-positive Early-stage Breast Cancer Management
Acronym: HERCard
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network); Ospedale Di Summa-Perrino (Unknown)
Responsible Party: Sponsor
Other Study IDs: INT 138/24
Record Dates: First submitted 2024-12-20; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3); HER2
Keywords: HER2-positive; operable breast cancer; gene-expression based classifier; prognosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Tumor tissue RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess the prognostic value of a genomic classifier (S18) and its refined version (S*) in women with early-stage HER2-positive breast cancer. The study aims to determine whether these tools can predict event-free (EFS) and disease-free survival (DFS) in patients treated with neoadjuvant and/or adjuvant trastuzumab-based therapies.

DETAILED DESCRIPTION:
The population includes women aged 18 or older with stage I-III HER2-positive breast cancer who received trastuzumab ± pertuzumab. Data and tumor tissue samples from this population have been collected prospectively from Istituto Nazionale dei Tumori IRCCS Fondazione Pascale, Naples (cohort A), and from Ospedale "Di Summa-Perrino", Brindisi (cohort B). The study integrates clinical-pathological and genomic data to refine and validate the prognostic capabilities of the S18 classifier.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Operable breast cancer (stage I-III)
3. Any status of hormone receptor in the primary tumor, according to institutional guidelines
4. HER2-positive primary tumor, according to ASCO guidelines, i.e., HER2-positive phenotype by immunohistochemistry (IHC) 3+ or 2+ with a positive result for ERBB2 gene amplification analysis using ISH techniques (CISH, SISH, FISH)
5. Neoadjuvant and/or adjuvant therapy based on trastuzumab ± pertuzumab
6. Written informed consent from patients

Exclusion Criteria:

1. Patient in follow-up for less than 3 years after surgery
2. A prior diagnosis of invasive cancer before the diagnosis of breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical information and paraffin-embedded tumor tissue samples from HER2-positive operable breast cancer patients included in the study were prospectively and consecutively collected at the participating centers and are now being analyzed for the purpose of the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) and Disease-free survival (DFS) according to the value of S18 and S* | From the initiation of systemic therapy through to at least 3 years post-treatment.
  To assess the prognostic value of the gene expression based classifier, with or without the integration of clinical-pathological variables, in patients receiving neoadjuvant and/or adjuvant chemotherapy with trastuzumab ± pertuzumab, with respect to event-free survival (EFS) and disease-free survival (DFS).

SECONDARY OUTCOMES:
Explorative evaluation of overall survival (OS) according to the value of S18 and S* | From the initiation of therapy through to at least 3 years post-treatment.
  To assess the prognostic value of the gene expression based classifier, with or without the integration of clinical-pathological variables, in patients receiving neoadjuvant and/or adjuvant chemotherapy with trastuzumab ± pertuzumab, with respect to overall survival (OS).
Evaluation of pathological complete response (pCR) according to the value of S18 and S* | Assessed in the surgical specimen obtained from definitive surgery performed within up to 10 months of initiating neoadjuvant treatment.
  To evaluate the predictive value of the gene expression based classifier in relation to pathological complete response (i.e., absence of breast cancer cells in surgical specimens) following neoadjuvant therapy with chemotherapy plus trastuzumab ± pertuzumab.

CONTACTS AND LOCATIONS:
Overall Officials: Serena Di Cosimo, MD, PhD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano; Paolo Verderio, PhD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano
Locations (2):
- Italy (2):
  - Ospedale Di Summa-Perrino, Brindisi
  - Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale, Naples

IPD SHARING:
Plan to Share IPD: Undecided
Our best efforts will be made to make IPD available in accordance with privacy, data security, and compliance with legal and ethical standards in place at the time of the study's conclusion. As of now, while the sharing of IPD remains a goal, these factors may occasionally present challenges that will need to be carefully addressed to ensure all necessary protections are in place at the appropriate time.